CLINICAL TRIAL: NCT06335914
Title: Dual PSMA and FDG PET Imaging for Patients With Advanced Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: dualPET-mPC; CAPCR: 23-5595 (Other: University Health Network)
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Advanced Prostate Cancer
Keywords: Prostate Specific Membrane Antigen; Positron Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PSMA and FDG PET Imaging (Experimental): Participants advanced prostate cancer will undergo PSMA and FDG PET prior to starting their standard of care treatment and during treatment.
  Interventions: Diagnostic Test: Ga 68 PSMA-11 PET; Diagnostic Test: 18F-DCFPyL PET; Diagnostic Test: FDG PET

INTERVENTIONS:
Diagnostic Test: Ga 68 PSMA-11 PET — Positron emission tomography (PET) imaging using Ga68 PSMA 11 radiotracer
Diagnostic Test: 18F-DCFPyL PET — Positron emission tomography (PET) imaging using 18F-DCFPyL radiotracer.
Diagnostic Test: FDG PET — Positron emission tomography (PET) imaging using (18) F-fluorodeoxyglucose radiotracer.

SUMMARY:
This study will use Prostate Specific Membrane Antigen (PSMA) and (18)F-Fluorodeoxyglucose Positron Emission Tomography (FDG PET) imaging in patients with advanced prostate cancer to learn about tumor biology across disease stages and during treatment. This may help with treatment selection and potential response monitoring in the future.

ELIGIBILITY:
Inclusion Criteria:

* Male, age ≥ 18 years
* Histologically or cytologically confirmed prostate cancer (adenocarcinoma)
* Poor risk patients with mCSPC at study enrollment
* De novo or recurrent high volume mCSPC as per conventional imaging (CT chest abdomen pelvis, or MRI, plus bone scan) prior to starting ADT and ARPI
* High or low volume mCSPC plus PSA ≥4.0 after 6-8 months of initiating ADT
* Willing to undergo study PET scans and remain under the care of medical oncology, radiation oncology or urology physician at Princess Margaret Cancer Center.
* No prior PSMA or FDG PET imaging within the last 60 days at each specified time point on study
* Patients enrolled in clinical trials are eligible if they satisfy all other criteria of eligibility

Exclusion Criteria:

* Under a randomized-controlled trial with unknown allocation of systemic therapy
* Inability to undergo or successfully complete PSMA PET and FDG PET imaging exams
* Unable to provide written consent by patient and their legal representatives
* In the opinion of the treating physician:
* conditions which would significantly impair the patient's ability to comply with study procedures and follow up
* Significant uncontrolled comorbidity, which may negatively impact the safety or interpretability of study PET imaging

  * another active malignancy
  * patient on dialysis
  * another radioisotope or investigational systemic agent within 5 half-lives prior to PET imaging

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2029-03-04 (Estimated); Study Completion 2029-09-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with high volume mCSPC having PSMA avid disease | 5 years

SECONDARY OUTCOMES:
Proportion of patients with PSMA-/FDG+ discordant lesions | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Di (Maria) Jiang, Principal Investigator — Princess Margaret Cancer Centre/University Health Network
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No